CLINICAL TRIAL: NCT01111175
Title: Triple Negative Breast Cancer Biomarker Study
Status: Completed | Type: Observational
Sponsor: US Oncology Research (Industry)
Collaborators: Translational Drug Development (Other); Life Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-133
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Breast Cancer; Triple Negative Breast Cancer
Keywords: Locally recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tumor tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with metastatic or locally recurrent triple negative breast cancer (TNBC) who are scheduled for medically indicated surgical biopsy or resection of disease will be identified. Fresh/frozen tissue will be collected and will undergo comprehensive molecular evaluation with NextGen sequencing. TGEN's clonal genomics analyses will be applied in the analysis to identify and prioritize the mutated targets. Therapeutic options, based on the genetic profile of each patient's tumor, will be discussed and an appropriate molecularly-selected agent will be recommended by the Study Investigator(s) (SI) and treating oncologist as treatment for the patient.

This is an open-label, pilot trial. Patients with metastatic or locally recurrent TNBC who are scheduled for medically indicated surgical biopsy or resection will be enrolled and therapeutic options, based on the genetic profile of each patient's tumor, will be discussed with the patient.

Time-to-progression (TTP) for these patients following the selected therapy is the primary objective and will be compared to the TTP(s) for their most recent prior therapy. A 30% increase in TTP with the molecularly-targeted agent compared with the TTP on the immediate prior therapy will be considered as evidence of clinical benefit from the selected therapy. The secondary endpoints are best response to the molecularly-selected therapy, overall survival (OS) and genetic mutation evaluation in metastatic (or locally recurrent) TNBC.

The study is designed to demonstrate that the collection and analysis of these tumor samples is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Has metastatic or locally recurrent triple negative breast cancer and is scheduled for medically indicated surgical biopsy or resection of disease
* Will have measurable or evaluable (nonmeasurable) disease per RECIST v 1.1 (see Section 10) present after surgical biopsy/resection. Note: following surgical resection, if the tumor sample is found to be inadequate for comprehensive molecular analysis, the patient will be deemed ineligible and will be replaced.
* Has received at least 1 prior chemotherapeutic regimen for their metastatic or locally recurrent TNBC prior to initiating the molecularly-selected therapy. There is no limit on the prior therapy for TNBC. Note: We strongly recommend holding of on intervening therapy if possible from the time of biopsy to the completion of sequencing so as not to change the cancer under the selective pressure of treatment, so that the sequencing results are reflective of the current cancer.
* Is at least 18 years of age
* Has an expected survival of at least 6 months, as estimated by the treating oncologist
* Has planned surgical resection (indicated for the medical care of the patient) that will yield a minimum fresh/frozen tumor sample of 1 cm x 1 cm x 1 cm (~300 mg) that will be available for molecular profiling analysis.
* Is agreeable to having a blood sample (10-20 mL) drawn and analyzed to compare their normal genetic profile to that of their tumor sample
* Has signed the most recent Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

* Has breast cancer other than metastatic or locally recurrent TNBC. Note: surgical resection of the recurrent TNBC will render the patient as "no evidence of disease" (NED). NED patients are ineligible and will be replaced.
* Has a history of heart disease, other conditions that would prevent treatment with a standard chemotherapeutic agent
* Has evidence of central nervous system (CNS) involvement that is progressing or that requires radiation, resection or steroid therapy
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
* Is a pregnant or nursing woman
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Evaluable patients with metastatic or locally advanced TNBC who are scheduled for surgical tumor biopsy or resection
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Time-to-progression (TTP) | Throughout study, for up to 3 years
  Time-to-progression (TTP) for these patients following the selected therapy is the primary objective and will be compared to the TTP(s) for their most recent prior therapy.

SECONDARY OUTCOMES:
Best response | To molecularly selected therapy, for up to 3 years
  Best response to therapy selected based on genomic analysis will be determined. Response will be evaluated in this study using the international criteria published by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee v1.1.
Overall survival | Throughout the study, for up to 3 years
  Survival will be measured, from the selected treatment start date to the date of death or the last date the patient was known to be alive.
Genetic mutation evaluation | After surgical resection
  Genomic analysis of whole blood and resected tumor will be done

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A O'Shaughnessy, MD, Principal Investigator — US Oncology Research; Daniel Von Hoff, MD, Principal Investigator — Translational Drug Development; John Carpten, PhD, Principal Investigator — Translational Drug Development
Locations (15):
- United States (15):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Virginia Oncology Assocites, Elizabeth City, North Carolina
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Oncology Associates, Williamsburg, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington